CLINICAL TRIAL: NCT03369730
Title: Early Stage Identification and Engagement to Reduce Duration of Untreated Psychosis (EaSIE)
Brief Title: Reducing the Duration of Untreated Psychosis in the United States
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yulia Landa, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-0655; R34MH115463 (NIH)
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: First Episode Psychosis (FEP); At Risk Mental State (ARMS)
Keywords: Screening; Duration of Untreated Psychosis (DUP); Coordinated Specialty Care (CSC); First Episode Psychosis (FEP); At Risk Mental State (ARMS); Clinical High Risk for Psychosis (CHR)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this project is to investigate whether a systematic screening approach for individuals with first episode psychosis (FEP) can substantially reduce Duration of Untreated Psychosis (DUP). The study team will evaluate the feasibility of screening a consecutive help-seeking population entering mental health services in order to facilitate early identification of FEP cases, rapid referral to specialty care and engagement in treatment.

DETAILED DESCRIPTION:
Psychosis typically emerges in late adolescence or early adulthood, during a vital stage in social and cognitive development, which can have a profoundly adverse impact on an individual's long-term functioning. Numerous studies find a substantial delay between the onset of psychosis and the initiation of specialty treatment for first episode psychosis (FEP), with the duration of untreated psychosis (DUP) typically over one year in the U.S. Better detection strategies are needed to improve identification of individuals with FEP and to rapidly engage them in Coordinated Specialty Care (CSC) aimed at restoring functioning. The onset of psychosis is preceded by a prodromal phase characterized by attenuated psychotic symptoms and decline in functioning. This phase (at-risk mental state: ARMS) is a potential target for strategies aimed at improving outcome by reducing DUP through regular symptom monitoring. This study will investigate whether a U.S. adaptation of a successful detection approach from the Netherlands can reduce DUP in the U.S. setting. The Dutch study found that screening of a consecutive help-seeking population entering mental health services captures significantly more FEP and ARMS cases than clinician referrals from mental health centers. Therefore screening may be an effective strategy for identifying individuals with psychotic symptoms earlier on in the course of their illness. This study will implement and evaluate a systematic screening for psychotic symptoms in community mental health clinics in order to facilitate rapid identification and engagement in treatment of individuals with FEP. Individuals ages 12 to 30 entering child/adolescent and adult community mental health clinics (CMHCs) within Mount Sinai Health System will be screened with the Prodromal Questionnaire - Brief Version (PQ-B). Those who screen positive will be assessed by the Structured Interview for Prodromal Syndromes (SIPS) and referred to stage-specific specialty care. Individuals with FEP will be referred to CSC programs: OnTrackNY and PEER. Individuals with ARMS will be monitored and referred to ICanFeelBetter program for ARMS. DUP will be measured for all individuals who meet SIPS psychosis criteria. The study team hypothesizes that screening for psychotic symptoms in CMHCs will be feasible and acceptable, and that the average DUP of FEP individuals identified with screening will be less than 3 months, the maximum time between onset of psychotic symptoms and engagement in CSC recommended by the World Health Organization. In order to optimize screening and treatment engagement strategies for reducing DUP, the clinical team will identify facilitators and barriers to FEP care through in-depth qualitative interviews with patients and caregivers, and by mapping pathways to FEP care. The study team will also conduct in-depth qualitative interviews with clinicians to explore their experience with the screening and referral process.

ELIGIBILITY:
Inclusion Criteria:

* age 12- 30
* ability to participate in assessments in English
* ability to provide informed consent (assent for those under age 18)
* meet criteria for psychosis or psychosis risk on SIPS

Exclusion Criteria:

* previous diagnosis of schizophrenia or schizoaffective disorder.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals ages 12 to 30 entering child/adolescent and adult community mental health clinics.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Duration of Untreated Psychosis (DUP) | Day 1
  The DUP is defined as the time, in weeks, between onset of psychotic symptoms and initiation of FEP treatment, in the case of this study, entry into Coordinated Specialty Care (CSC) programs for first episode psychosis (FEP).

SECONDARY OUTCOMES:
Rate of completed PQ-B screen. | Day 1
  Rate of completed Prodromal Questionnaire - Brief Version (PQ-B) of incoming patients in clinics. Screen given as part of standard care. The PQ-B is a 21-item screening measure used to predict classification of psychosis or psychosis-risk on the Structured Interview for Psychosis-risk Syndromes (SIPS).
Rate of completed SIPS | Day 1
  Rate of completed Interview for Psychosis-risk Syndromes (SIPS) of incoming patients in clinics. Screen given as part of standard care. SIPS is a structured interview for diagnosing a clinical high risk (CHR) syndrome for psychosis and cases of first episode psychosis (FEP).
Rates of FEP cases | Day 1
  Rates of (First Episode Psychosis) FEP cases detected
Rate of ARMS cases | Day 1
  Rate of At Risk Mental State (ARMS) cases detected
Rate of CHR cases | Day 1
  Rate of Clinical High Risk for Psychosis (CHR) cases detected

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Landa, PsyD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Trustees of Boston University, Boston, Massachusetts
  - Research Foundation/City University of New York (CUNY) on behalf of CUNY Graduate School, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
In accordance with NIH policy, a de-identified dataset will be uploaded to the NIMH Data Archive: the National Database for Clinical Trials Related to Mental Illness.

REFERENCES:
- [Background] Addington J, Heinssen RK, Robinson DG, Schooler NR, Marcy P, Brunette MF, Correll CU, Estroff S, Mueser KT, Penn D, Robinson JA, Rosenheck RA, Azrin ST, Goldstein AB, Severe J, Kane JM. Duration of Untreated Psychosis in Community Treatment Settings in the United States. Psychiatr Serv. 2015 Jul;66(7):753-6. doi: 10.1176/appi.ps.201400124. Epub 2015 Jan 15. PMID 25588418
- [Background] Dixon LB, Goldman HH, Bennett ME, Wang Y, McNamara KA, Mendon SJ, Goldstein AB, Choi CW, Lee RJ, Lieberman JA, Essock SM. Implementing Coordinated Specialty Care for Early Psychosis: The RAISE Connection Program. Psychiatr Serv. 2015 Jul;66(7):691-8. doi: 10.1176/appi.ps.201400281. Epub 2015 Mar 16. PMID 25772764
- [Background] Rietdijk J, Klaassen R, Ising H, Dragt S, Nieman DH, van de Kamp J, Cuijpers P, Linszen D, van der Gaag M. Detection of people at risk of developing a first psychosis: comparison of two recruitment strategies. Acta Psychiatr Scand. 2012 Jul;126(1):21-30. doi: 10.1111/j.1600-0447.2012.01839.x. Epub 2012 Feb 15. PMID 22335365